CLINICAL TRIAL: NCT05582213
Title: Effect of Ketamine Versus Sevoflurane On The Right Ventricular Pressure During Congenital Pulmonary Stenosis Balloon Dilatation
Brief Title: Effect of Ketamine Versus Sevoflurane On The Right Ventricular Pressure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amr Gaber, lecturer clinical doctor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: congenital pulmonary stenosis
Record Dates: First submitted 2022-10-10; First posted 2022-10-17 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Congenital Pulmonary Stenosis
MeSH Terms: conditions — Stenosis, Pulmonary Artery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- classic group (CL group) (Other): 20 patients will be enrolled to induction with sevofloran as inhalational anesthetics
  Interventions: Diagnostic Test: induction of anesthesia
- Group ketamine: (Other): This group includes (20) patients will receive ketamine 2 mg/kg intravenous for induction of sedation and unconsciousness
  Interventions: Diagnostic Test: induction of anesthesia

INTERVENTIONS:
Diagnostic Test: induction of anesthesia — This group includes (20) patients will receive induction by sevoflurane 3% using open circuit (modified Ayre's T-piece) till loss of consciousness and will be maintained on oxygen mask on the same concentration of sevoflurane and connected to capnogram

SUMMARY:
The aim of this study is to compare the effect of different anesthetic drugs used for induction of anesthesia ketamine versus sevoflurane on the RV pressure in pediatrics undergoing balloon dilatation for congenital pulmonary stenosis.

DETAILED DESCRIPTION:
Critical pulmonary stenosis (PS) is a life-threatening congenital heart disease which manifest during the neonatal period with cyanosis. Surgical valvotomy was the procedure of choice for critical PS; however, balloon pulmonary valvoplasty (BPV) has now become the standard management.

Ketamine is often used for procedural sedation or as adjunct agent for general anesthesia in pediatrics with congenital heart disease. Ketamine is a chemical derivative of phencyclidine acting as a selective antagonist of the N-methyl-d-aspartate (NMDA) receptor, an ionotropic glutamate receptor that participates in analgesia, amnesia, and sedation pathways.

Ketamine has minimal impact on hemodynamics in children with congenital heart disease when used at usual clinical doses. Systemic vascular resistance and pulmonary vascular resistance are not significantly altered.

Sevoflurane is a sweet-smelling, highly fluorinated methyl isopropyl ether used as an inhalational anesthetic for induction and maintenance of general anesthesia. It proved to be safe as induction agent in noncardiac surgery and cardiac surgery. Sevoflurane has low solubility in blood, produces less arrhythmias and decrease in contractility less than halothane without changing pulmonary to systemic blood flow ratio in pediatrics with congenital heart disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 1 month to 1 year.
2. Both gender
3. Isolated congenital pulmonary stenosis

Exclusion Criteria:

1. Multiple cardiac congenital anomalies.
2. Previous open-heart surgery.
3. Other non-cardiac congenital anomalies
4. Refusal of parents

Ages: 1 Month to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-10 (Actual)

PRIMARY OUTCOMES:
right ventricular pressure | baseline
  right ventricular pressure before induction of anesthesia

SECONDARY OUTCOMES:
vital data | baseline
  Spo2 in both group

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

REFERENCES:
- [Background] Hoetama E, Prakoso R, Roebiono PS, Sakidjan I, Kurniawati Y, Siagian SN, Lelya O, Rahajoe AU, Harimurti GM, Lilyasari O. Balloon pulmonary valvuloplasty in neonates with critical pulmonary stenosis: Jugular or femoral. Ann Pediatr Cardiol. 2020 Jan-Mar;13(1):11-15. doi: 10.4103/apc.APC_14_19. Epub 2019 Nov 7. PMID 32030030
- [Background] Loomba RS, Gray SB, Flores S. Hemodynamic effects of ketamine in children with congenital heart disease and/or pulmonary hypertension. Congenit Heart Dis. 2018 Sep;13(5):646-654. doi: 10.1111/chd.12662. Epub 2018 Sep 27. PMID 30259660
- [Background] Sungur Ulke Z, Kartal U, Orhan Sungur M, Camci E, Tugrul M. Comparison of sevoflurane and ketamine for anesthetic induction in children with congenital heart disease. Paediatr Anaesth. 2008 Aug;18(8):715-21. doi: 10.1111/j.1460-9592.2008.02637.x. PMID 18544145
- [Background] de Waard-van der Spek FB, van den Berg GM, Oranje AP. EMLA cream: an improved local anesthetic. Review of current literature. Pediatr Dermatol. 1992 Jun;9(2):126-31. doi: 10.1111/j.1525-1470.1992.tb01228.x. No abstract available. PMID 1603740
- [Background] Herregods L, Mortier E, Donadoni R, Rolly G. A comparison of midazolam and diazepam for sedation during locoregional anesthesia. Acta Anaesthesiol Belg. 1987;38(1):97-102. PMID 3591272
- [Background] Berkenbosch JW, Wankum PC, Tobias JD. Prospective evaluation of dexmedetomidine for noninvasive procedural sedation in children. Pediatr Crit Care Med. 2005 Jul;6(4):435-9; quiz 440. doi: 10.1097/01.PCC.0000163680.50087.93. PMID 15982430
- [Background] Furyk JS, Meek RA, Egerton-Warburton D. Drugs for the treatment of nausea and vomiting in adults in the emergency department setting. Cochrane Database Syst Rev. 2015 Sep 28;2015(9):CD010106. doi: 10.1002/14651858.CD010106.pub2. PMID 26411330
- [Background] 8. Eric Scholar, in xPharm: The Comprehensive Pharmacology Reference, 2007
- [Background] Williams GD, Philip BM, Chu LF, Boltz MG, Kamra K, Terwey H, Hammer GB, Perry SB, Feinstein JA, Ramamoorthy C. Ketamine does not increase pulmonary vascular resistance in children with pulmonary hypertension undergoing sevoflurane anesthesia and spontaneous ventilation. Anesth Analg. 2007 Dec;105(6):1578-84, table of contents. doi: 10.1213/01.ane.0000287656.29064.89. PMID 18042853
- [Background] Meyers RS. Pediatric fluid and electrolyte therapy. J Pediatr Pharmacol Ther. 2009 Oct;14(4):204-11. doi: 10.5863/1551-6776-14.4.204. PMID 23055905
- [Background] 11. Rajan S, Tosh P, Sudevan M, Rahman AA, Kumar L. Anaesthetic management of a child with tetralogy of Fallot for dental extraction: a modified technique. Research and Opinion in Anesthesia and Intensive Care. 2019 Oct 1;6(4):470.
- [Background] Russell IA, Miller Hance WC, Gregory G, Balea MC, Cassorla L, DeSilva A, Hickey RF, Reynolds LM, Rouine-Rapp K, Hanley FL, Reddy VM, Cahalan MK. The safety and efficacy of sevoflurane anesthesia in infants and children with congenital heart disease. Anesth Analg. 2001 May;92(5):1152-8. doi: 10.1097/00000539-200105000-00014. PMID 11323338